CLINICAL TRIAL: NCT01380990
Title: Phase I/II, Historical Controlled, Open-label, Non-randomised, Single-centre Trial to Assess the Safety and Efficacy of EF1αS-ADA Lentiviral Vector Mediated Gene Modification of Autologous CD34+ Cells From ADA-deficient Individuals
Brief Title: Lentiviral (LV) Gene Therapy for Adenosine Deaminase (ADA) Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Orchard Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-MI-29
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Adenosine Deaminase Deficiency; Severe Combined Immunodeficiencies (SCID)
Keywords: Gene therapy; Hematopoietic stem and progenitor cells; Lentiviral vector; ADA-SCID
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Severe Combined Immunodeficiency | interventions — Busulfan; pegademase bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gene Therapy (Experimental): Infusion of autologous EFS-ADA LV CD34+ cells
  Interventions: Genetic: Infusion of autologous EFS-ADA LV CD34+ cells; Drug: Busulfan; Drug: Peg-Ada
- Historical Control Group (Other): Historical data from ADA-SCID patients who were treated with Hematopoietic Stem Cell Transplantation (HSCT)
  Interventions: Other: Haematopoietic Stem Cell Transplantation (HSCT)

INTERVENTIONS:
Genetic: Infusion of autologous EFS-ADA LV CD34+ cells — Autologous EFS-ADA LV CD34+ cells (OTL-101*) are infused intravenously
  Other Names: OTL-101*
  Arms: Gene Therapy
Other: Haematopoietic Stem Cell Transplantation (HSCT) — Historical data from a database of ADA-SCID patients treated with allogeneic HSCT from GOSH will be collected as comparator group.
  Arms: Historical Control Group
Drug: Busulfan — Busulfan is used for non-myeloablative conditioning
  Arms: Gene Therapy
Drug: Peg-Ada — Peg-Ada enzyme replacement therapy is discontinued at Day +3- (-3/+15 days) after successful engraftment
  Arms: Gene Therapy

SUMMARY:
This is a historically controlled, non-randomized Phase I/II clinical trial to assess the safety and efficacy of autologous transplantation of CD34+ hematopoietic stem/progenitor cells (HSPCs), obtained from infants affected by ADA-SCID, following transduction of the HSPCs with a lentiviral vector (LV) carrying the human ADA complementary DNA (cDNA) under the control of the elongation factor 1 alpha shortened (EFS) promoter. Subjects treated in the trial receive the infusion of autologous, transduced cells following marrow cytoreduction with busulfan. The outcomes are compared to those observed in a historical control group of patients who received an allogeneic hematopoietic stem cell transplant (HSCT).

This Phase I/II clinical trial will be performed at Great Ormond Street Hospital (GOSH), London, United Kingdom.

ELIGIBILITY:
Gene Therapy (On Trial)

Inclusion Criteria:

1. Diagnosis of ADA-SCID confirmed by DNA sequencing or by confirmed absence of <3% of ADA enzymatic activity in peripheral blood (or for neonates) in umbilical cord blood erythrocytes and/or leukocytes or in cultured fetal cells derived from either chorionic villus biopsy or amniocentesis, prior to institution of Polyethylene glycol-modified ADA (PEG-ADA) replacement therapy
2. Patients who lack a fully Human leukocyte antigen (HLA)-matched family donor
3. Patients (male or female) <5 years of age OR Patients (male or female) ≥ 5 years to 15 years of age who have preserved thymic function as evidenced by presence of >10 % naïve T cells (CD4+45RA+27+ cells)
4. Parental/guardian signed informed consent

Exclusion Criteria:

1. Cytogenetic abnormalities on peripheral blood
2. Evidence of active malignant disease
3. Known sensitivity to busulfan
4. If applicable, confirmed pregnancy (to be tested in patients above 12 years old)

Gene Therapy (CUP)

A group of patients were treated under CUP (GOSH special license) either because the study was not yet open and patients needed urgent treatment, or because they were outside of the inclusion/exclusion criteria or received Investigational Medicinal Product (IMP) followed a different process (ie, received in two infusions). Patients followed the same protocol steps and study visits.

Historical Control Group

Inclusion Criteria:

1. Diagnosis of ADA-SCID confirmed by DNA sequencing OR by confirmed absence of <3% of ADA enzymatic activity in peripheral blood or (for neonates) in umbilical cord blood erythrocytes and/or leucocytes or in cultured foetal cells derived from either chorionic villus biopsy or amniocentesis, prior to institution of PEG-ADA replacement therapy
2. Patients (male or female) between 0-18 years at time of treatment
3. Patient treated with allogeneic haematopoietic stem cell transplantation since 2000

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2012-11-15 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Booth, Dr, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Kohn DB, Booth C, Shaw KL, Xu-Bayford J, Garabedian E, Trevisan V, Carbonaro-Sarracino DA, Soni K, Terrazas D, Snell K, Ikeda A, Leon-Rico D, Moore TB, Buckland KF, Shah AJ, Gilmour KC, De Oliveira S, Rivat C, Crooks GM, Izotova N, Tse J, Adams S, Shupien S, Ricketts H, Davila A, Uzowuru C, Icreverzi A, Barman P, Campo Fernandez B, Hollis RP, Coronel M, Yu A, Chun KM, Casas CE, Zhang R, Arduini S, Lynn F, Kudari M, Spezzi A, Zahn M, Heimke R, Labik I, Parrott R, Buckley RH, Reeves L, Cornetta K, Sokolic R, Hershfield M, Schmidt M, Candotti F, Malech HL, Thrasher AJ, Gaspar HB. Autologous Ex Vivo Lentiviral Gene Therapy for Adenosine Deaminase Deficiency. N Engl J Med. 2021 May 27;384(21):2002-2013. doi: 10.1056/NEJMoa2027675. Epub 2021 May 11. PMID 33974366

RESULTS

PARTICIPANT FLOW:
Groups:
- Gene Therapy: Infusion of autologous EF1αS-ADA (EFS-ADA) lentiviral vector (LV) mediated gene modification of autologous CD34+ cells
  Infusion of autologous EFS-ADA LV CD34+ cells: Autologous EFS-ADA LV CD34+ cells (OTL-101*) are infused intravenously
  Busulfan: Busulfan is used for non-myeloablative conditioning
  Polyethylene glycol-modified adenosine deaminase (PEG-ADA): PEG-ADA enzyme replacement therapy (ERT) is discontinued at Day +3- (-3/+15 days) after successful engraftment
- Historical Control Group: Historical data from patients with Severe Combined Immunodeficiency Due to ADA Deficiency (ADA-SCID) who were treated with Hematopoietic Stem Cell Transplantation (HSCT)
  Haematopoietic Stem Cell Transplantation (HSCT): Historical data from a database of ADA-SCID patients treated with allogeneic HSCT from Great Ormond Street Hospital (GOSH) will be collected as comparator group.
Period: Overall Study
Arm/Group | Gene Therapy | Historical Control Group
Started | 20 | 16
Completed | 19 | 15
Not Completed | 1 | 1
Not completed — Treatment Failure | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants were included in the Baseline Analysis Population
Groups:
- Gene Therapy: The safety population consists of all OTL-101*-treated subjects (on-study and CUP). The secondary efficacy population consists of all OTL-101*-treated subjects (on-study and CUP).
- Historical Control Group: Complete HSCT historical control group consisting of ADA-SCID patients with any type of donor treated with HSCT at GOSH from 2000 to 2016 (referred to as the All HSCT Controls group)
- Total: Total of all reporting groups
Arm/Group | Gene Therapy | Historical Control Group | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 16 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex, n: Female | 8 | 0 | 8
  Sex, n: Male | 12 | 0 | 12
  Sex, n: Not Reported | 0 | 16 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity, n: Asian | 2 | 0 | 2
  Ethnicity, n: White European | 10 | 0 | 10
  Ethnicity, n: Other | 6 | 0 | 6
  Ethnicity, n: Unknown | 2 | 0 | 2
  Ethnicity, n: Not reported | 0 | 16 | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Subjects Treated With Investigational Medicinal Product (IMP) (1 Year)
Description: Overall survival is defined as the percentage of subjects alive at 12 months post- treatment with OTL-101* or HSCT
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- OTL-101* On-Study Subjects: The primary efficacy population for analysis consists of the on-study OTL-101*-treated subjects.
- OTL-101* On-Study and CUP Subjects: The safety population consists of all OTL-101*-treated subjects (on-study and CUP). The secondary efficacy population consists of all OTL-101*-treated subjects (on-study and CUP).
- HSCT Controls Without MRD: The primary efficacy population from the HSCT historical control cohort comprises ADA-SCID patients without a medically eligible Matched Related Donor (MRD) who were treated with HSCT at GOSH from 2000 to 2016. An MRD refers to either a matched sibling or family donor.
- HSCT Controls With MRD: Secondary efficacy population for comparison comprise ADA-SCID patients with an MRD treated with HSCT at GOSH from 2000 to 2016
- All HSCT Controls: Complete HSCT historical control group consisting of ADA-SCID patients with any type of donor treated with HSCT at GOSH from 2000 to 2016 (referred to as the All HSCT Controls group)
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 10 | 20 | 5 | 11 | 16
percentage of participants | 100 [69.15 to 100] | 100 [83.16 to 100] | 100 [47.82 to 100] | 100 [71.51 to 100] | 100 [79.41 to 100]
Statistical Analysis 1: Comparison: OTL-101* On-Study Subjects vs HSCT Controls Without MRD; Percentage of patients alive at 1-year post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients alive at 1-year post-treatment with OTL-101* (on-study). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 2: Comparison: OTL-101* On-Study Subjects vs HSCT Controls With MRD; Percentage of patients alive at 1-year post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients alive at 1-year post-treatment with OTL-101* (on-study). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 3: Comparison: OTL-101* On-Study Subjects vs All HSCT Controls; Percentage of patients alive at 1-year post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients alive at 1-year post-treatment with OTL-101* (on-study). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 4: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls Without MRD; Percentage of patients alive at 1-year post-treatment in the historical control groups (without MRD) were compared to the percentage of patients alive at 1-year post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 5: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls With MRD; Percentage of patients alive at 1-year post-treatment in the historical control groups (with MRD) were compared to the percentage of patients alive at 1-year post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 6: Comparison: OTL-101* On-Study and CUP Subjects vs All HSCT Controls; Percentage of patients alive at 1-year post-treatment in the historical control groups (all historical controls) were compared to the percentage of patients alive at 1-year post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0

2. Primary Outcome: Event-free Survival (EvFS) of Subjects Treated With Investigational Medicinal Product (IMP) (1 Year)
Description: Event-free survival is defined as the percentage of subjects alive with no "event", an "event" being the resumption of PEG-ADA ERT or the need for a rescue allogenic Hematopoietic Stem Cell Transplant (HSCT), or death.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HSCT Controls Without MRD: The primary efficacy population from the HSCT historical control cohort comprises ADA-SCID patients without a medically eligible MRD who were treated with HSCT at GOSH from 2000 to 2016. An MRD refers to either a matched sibling or family donor.
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 10 | 20 | 5 | 11 | 16
percentage of participants | 100 [69.15 to 100] | 100 [83.16 to 100] | 100 [47.82 to 100] | 100 [71.51 to 100] | 100 [79.41 to 100]
Statistical Analysis 1: Comparison: OTL-101* On-Study Subjects vs HSCT Controls Without MRD; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101* (on-study). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 2: Comparison: OTL-101* On-Study Subjects vs HSCT Controls With MRD; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101* (on-study). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 3: Comparison: OTL-101* On-Study Subjects vs All HSCT Controls; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101* (on-study). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 4: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls Without MRD; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 5: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls With MRD; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 6: Comparison: OTL-101* On-Study and CUP Subjects vs All HSCT Controls; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0

3. Primary Outcome: Vector Copy Number (VCN) in Granulocytes Fraction (Neutrophils)
Description: Engraftment of transduced cells was assessed using vector gene marking in granulocytes (neutrophils)
Time Frame: 36 months
Population: Historical control groups/arms are not included in the analysis population for this outcome measure as these subjects did not receive gene therapy, and so measurement of VCN levels is not relevant
Measure: Median (Full Range); unit: copies/cell
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 9 | 18
copies/cell | 0.240 [0.15 to 0.79] | 0.280 [0.03 to 1.60]

4. Primary Outcome: VCN in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Engraftment of transduced cells was assessed using vector gene marking in PBMCs
Time Frame: 36 months
Population: as for outcome 3
Measure: Median (Full Range); unit: copies/cell
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 9 | 18
copies/cell | 0.600 [0.20 to 1.67] | 0.625 [0.20 to 1.67]

5. Primary Outcome: VCN in CD3+ T Cells
Description: Engraftment of transduced cells was assessed using vector gene marking
Time Frame: 36 months
Population: as for outcome 3
Measure: Median (Full Range); unit: copies/cell
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 8 | 17
copies/cell | 1.065 [0.84 to 1.59] | 1.160 [0.30 to 4.61]

6. Primary Outcome: VCN in CD19+ B Cells
Description: Engraftment of transduced cells was assessed using vector gene marking in CD19+ B Cells
Time Frame: 36 months
Population: as for outcome 3
Measure: Median (Full Range); unit: copies/cell
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 9 | 17
copies/cell | 0.880 [0.68 to 1.77] | 1.190 [0.68 to 3.75]

7. Primary Outcome: Change From Baseline in CD3+ T Cell Counts (1 Year)
Description: Immune reconstitution was assessed by change in CD3+ T Cell counts over time.
Time Frame: 12 months
Population: Historical control groups/arms are not included in the analysis population for this outcome measure as CD3+ T cell count data was not collected due to the historical nature of the population
Measure: Geometric Mean (95% Confidence Interval); unit: 10e9 cells/L
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 8 | 17
10e9 cells/L | 3.58 [1.64 to 7.83] | 3.18 [1.98 to 5.10]
Statistical Analysis 1: Comparison: OTL-101* On-Study Subjects; Mixed-Effect Model Repeated Measure (MMRM) Analysis of Change from Baseline to Month 12 in Log-Transformed CD3+ T Cell count (OTL-101*) for "OTL-101* on-study subjects" group; Test type: Other — Model includes fixed effects for visit and Baseline, subject as random effect, with compound symmetry covariance structure. Observations with a value of 0 were imputed as 0.01. Model analyses log transformed data, so the adjusted mean refers to the geometric mean ratio between Month 12 and Baseline; p = 0.002, Mixed Models Analysis
Statistical Analysis 2: Comparison: OTL-101* On-Study and CUP Subjects; MMRM Analysis of Change from Baseline to Month 12 in Log-Transformed CD3+ T Cell count (OTL-101*) for "OTL-101* on-study and CUP subjects" group; Test type: Other — [test comment as in outcome 7, analysis 1]; p < 0.001, Mixed Models Analysis

8. Primary Outcome: Change From Baseline in CD3+ T Cell Counts (3 Years)
Description: Immune reconstitution was assessed by change in CD3+ T Cell counts over time.
Time Frame: 36 months
Population: as for outcome 7
Measure: Median (Full Range); unit: 10e9 cells/L
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 7 | 16
10e9 cells/L | 1.060 [0.59 to 1.47] | 1.090 [-0.49 to 1.47]

9. Primary Outcome: ADA Activity in Erythrocytes
Description: ADA enzyme activity was assessed as a measure of successful engraftment of genetically modified Hematopoietic stem progenitor cells (HSPCs), as it marks sustained gene expression from the normal ADA transgene.
Time Frame: 36 months
Measure: Median (Full Range); unit: nmol/h/mg
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 8 | 16 | 3 | 7 | 10
nmol/h/mg | 638.0 [220 to 3038] | 490.5 [27 to 3038] | 86.5 [39 to 115] | 1.0 [0 to 27] | 23.0 [0 to 115]

10. Primary Outcome: Reduction in Deoxyadenosine Triphosphate (dATP) in Erythrocytes
Description: Decreased dATP levels coincide with increased ADA enzyme activity, detoxification was used as a marker of correction of the defective ADA gene. The threshold for detoxification was <100 μmol/L.
Time Frame: 36 months
Measure: Median (Full Range); unit: umol/L
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 6 | 12 | 1 | 5 | 6
umol/L | 50.0 [50 to 50] | 50.0 [50 to 50] | 0.0 [0 to 0] | 114.0 [23 to 192] | 90.0 [0 to 192]

11. Primary Outcome: Frequency of Vector Integration Into Known Protooncogenes (3 Years)
Description: Vector Integration Site Analysis (VISA) allowed determination of the distribution of vector integration sites in each subject's genome, as well as the relative clonal abundance. VISA was to be considered abnormal for a subject if, in 2 or more instances during the course of follow-up, a single integration site was found to represent >30% of the total integration sites detected.
  There were no instances of clonal proliferation in the course of the 36 month follow-up for on-study and CUP subjects; hence, a detailed analysis of the frequency of clonal expansion associated with vector integration near proto-oncogenes was not generated.
Time Frame: 36 months
Population: Historical control groups/arms are not included in the analysis population for this outcome measure as these subjects did not receive gene therapy, and so measurement of VISA is not relevant
Measure: Number; unit: % of integration in known protooncogenes
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects
Number analyzed (Participants) | 10 | 20
% of integration in known protooncogenes | 0 | 0

12. Secondary Outcome: OS of Subjects Treated With IMP With Those of Patients Treated With Allogeneic HSCT (3 Years)
Description: Overall survival (OS) is defined as the percentage of subjects alive at 36 months post- treatment with OTL-101* or HSCT
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 10 | 20 | 5 | 11 | 16
percentage of participants | 100 [66.37 to 100] | 100 [82.35 to 100] | 100 [47.82 to 100] | 88.89 [51.75 to 99.72] | 92.86 [66.13 to 99.82]
Statistical Analysis 1: Comparison: OTL-101* On-Study Subjects vs HSCT Controls Without MRD; Percentage of patients with OS at 3-years post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with OS at 3-years post-treatment with OTL-101* (on study). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 2: Comparison: OTL-101* On-Study Subjects vs HSCT Controls With MRD; Percentage of patients with OS at 3-years post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with OS at 3-years post-treatment with OTL-101* (on study). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 11.11, 95% CI 2-sided [-22.41 to 48.25]
Statistical Analysis 3: Comparison: OTL-101* On-Study Subjects vs All HSCT Controls; Percentage of patients with OS at 3-years post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients with OS at 3-years post-treatment with OTL-101* (on study). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 7.14, 95% CI 2-sided [-28.10 to 34.23]
Statistical Analysis 4: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls Without MRD; Percentage of patients with OS at 3-years post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with OS at 3-years post-treatment with OTL-101* (on study and CUP). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 5: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls With MRD; Percentage of patients with OS at 3-years post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with OS at 3-years post-treatment with OTL-101* (on study and CUP). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 11.11, 95% CI 2-sided [-10.01 to 48.25]
Statistical Analysis 6: Comparison: OTL-101* On-Study and CUP Subjects vs All HSCT Controls; Percentage of patients with OS at 3-years post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients with OS at 3-years post-treatment with OTL-101* (on study and CUP). Results are reported as percentage difference in OS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 7.14, 95% CI 2-sided [-12.91 to 33.87]

13. Secondary Outcome: EvFS of Subjects Treated With IMP With Those of Patients Treated With Allogeneic HSCT (3 Years)
Description: as for outcome 2
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 10 | 20 | 5 | 11 | 16
percentage of participants | 90.00 [55.50 to 99.75] | 95.00 [75.13 to 99.87] | 80.00 [28.36 to 99.49] | 60.00 [26.24 to 87.84] | 66.67 [38.38 to 88.18]
Statistical Analysis 1: Comparison: OTL-101* On-Study Subjects vs HSCT Controls Without MRD; Test type: Superiority; p = 0.645, Log Rank
Statistical Analysis 2: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls Without MRD; Test type: Superiority; p = 0.299, Log Rank
Statistical Analysis 3: Comparison: OTL-101* On-Study Subjects vs HSCT Controls With MRD; Test type: Superiority; p = 0.2, Log Rank
Statistical Analysis 4: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls With MRD; Test type: Superiority; p = 0.028, Log Rank
Statistical Analysis 5: Comparison: OTL-101* On-Study Subjects vs All HSCT Controls; Test type: Superiority; p = 0.259, Log Rank
Statistical Analysis 6: Comparison: OTL-101* On-Study and CUP Subjects vs All HSCT Controls; Test type: Superiority; p = 0.044, Log Rank
Statistical Analysis 7: Comparison: OTL-101* On-Study Subjects vs HSCT Controls Without MRD; Percentage of patients with EvFS at 3-years post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with EvFS at 3-years post-treatment with OTL-101* (on-study). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 10.00, 95% CI 2-sided [-32.05 to 61.97]
Statistical Analysis 8: Comparison: OTL-101* On-Study Subjects vs HSCT Controls With MRD; Percentage of patients with EvFS at 3-years post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with EvFS at 3-years post treatment with OTL-101* (on-study). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 30.00, 95% CI 2-sided [-10.72 to 65.87]
Statistical Analysis 9: Comparison: OTL-101* On-Study Subjects vs All HSCT Controls; Percentage of patients with EvFS at 3-years post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients with EvFS at 3-years post-treatment with OTL-101* (on-study). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study subjects; Test type: Superiority; Difference in percentages = 23.33, 95% CI 2-sided [-15.24 to 54.59]
Statistical Analysis 10: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls Without MRD; Percentage of patients with EvFS at 3-years post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with EvFS at 3-years post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 15.00, 95% CI 2-sided [-13.70 to 63.54]
Statistical Analysis 11: Comparison: OTL-101* On-Study and CUP Subjects vs HSCT Controls With MRD; Percentage of patients with EvFS at 3-years post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with EvFS at 3-years post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 35.00, 95% CI 2-sided [2.29 to 68.45]
Statistical Analysis 12: Comparison: OTL-101* On-Study and CUP Subjects vs All HSCT Controls; Percentage of patients with EvFS at 3-years post-treatment in the historical control groups (all historical controls) were compared to the percentage of study patients with EvFS at 3-years post-treatment with OTL-101* (on-study and CUP). Results are reported as percentage difference in EvFS of historical control group from OTL-101* on-study and CUP subjects; Test type: Superiority; Difference in percentages = 28.33, 95% CI 2-sided [2.04 to 56.36]

14. Secondary Outcome: Infection Rate
Description: The infections of interest in this study were severe infections or opportunistic infectious episodes, defined as infections requiring hospitalization or prolonging hospitalization and/or documented infections by opportunistic pathogens.
Time Frame: 36 months
Measure: Number; unit: Infection rate per person per year
Arm/Group | OTL-101* On-Study Subjects | OTL-101* On-Study and CUP Subjects | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Controls
Number analyzed (Participants) | 10 | 20 | 5 | 11 | 16
Infection rate per person per year | 0.14 | 0.14 | 0.13 | 0.17 | 0.16

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of participant consent, approximately 1-month pre-treatment, up until 3-years post-treatment with OTL-101*
Description: Adverse events were reported for subjects treated with OTL-101*.
  Adverse event reporting is not applicable for the historical control arms (without MRD, with MRD, and all control patients) as this data was not collected due to the historical nature of the population.
Groups:
- OTL-101* On-Study and CUP Subjects: The safety population consists of all OTL-101*-treated subjects (on-study and CUP).
- OTL-101* On-Study Subjects: The safety population for analysis consists of the on-study OTL-101*-treated subjects.
Arm/Group | OTL-101* On-Study and CUP Subjects | OTL-101* On-Study Subjects
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 11/20 | 7/10
Other Adverse Events (participants affected / at risk) | 20/20 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTL-101* On-Study and CUP Subjects (N=20) | OTL-101* On-Study Subjects (N=10)
Pyrexia (General disorders) | 6 (8) | 5 (7)
Device related infection (Infections and infestations) | 1 (1) | 3 (4)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Transmission of an infectious agent via product (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 2 (3) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTL-101* On-Study and CUP Subjects (N=20) | OTL-101* On-Study Subjects (N=10)
Rhinitis (Infections and infestations) | 9 (15) | 5 (9)
Viral upper respiratory tract infection (Infections and infestations) | 7 (12) | 4 (7)
Otitis media (Infections and infestations) | 3 (4) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Metapneumovirus infection (Infections and infestations) | 2 (2) | 2 (2)
Viral rash (Infections and infestations) | 2 (2) | 2 (2)
Ear infection (Infections and infestations) | 2 (3) | 1 (2)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (13) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (15) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (Infections and infestations) | 9 (16) | 4 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (19) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (10) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Sapovirus test positive (Investigations) | 2 (3) | 1 (2)
Norovirus test positive (Investigations) | 4 (4) | 1 (1)
Adenovirus test positive (Investigations) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Enterococcus test positive (Investigations) | 2 (2) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (9) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Ocular hyperaemia (Eye disorders) | 2 (2) | 2 (2)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Tinea capitis (Infections and infestations) | 1 (1) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (2) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acinetobacter test positive (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 1 (1)
Morganella test positive (Investigations) | 1 (1) | 1 (1)
Aspiration bone marrow abnormal (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Chest x-ray abnormal (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0)
Epstein-Barr virus test positive (Investigations) | 1 (3) | 0 (0)
Human metapneumovirus test positive (Investigations) | 1 (1) | 0 (0)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0)
Respirovirus test positive (Investigations) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 1 (1)
Infusion site erythema (General disorders) | 1 (1) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 1 (1) | 1 (1)
Amblyopia (Eye disorders) | 1 (1) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Gross motor delay (Nervous system disorders) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Combined immunodeficiency (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Preauricular cyst (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT01380990/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT01380990/SAP_001.pdf